CLINICAL TRIAL: NCT04378920
Title: A Study of Liposomal Trans Crocetin, LEAF-4L6715, in Patients With Acute Respiratory Distress Syndrome Due to COVID-19, Sepsis or Other Causes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: LEAF4Life, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003; 2020-001393-30 (EudraCT Number); 2020-A00900-39 (Other: IDRCB)
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: COVID19, Sepsis or Other Causes; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Sepsis; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 4L6715 (Experimental): exploring various doses of LEAF-4L6715
  Interventions: Drug: LEAF-4L6715

INTERVENTIONS:
Drug: LEAF-4L6715 — LEAF-4L6715

SUMMARY:
This is an open label phase II study of treatment with LEAF-4L6715 in patients who experience severe acute respiratory distress syndrome (ARDS) due to COVID-19, Sepsis or other Causes. The purpose of this study is to evaluate the improvement in PaO2/FiO2 by more than 25% in patients treated with LEAF-4L6715.

DETAILED DESCRIPTION:
Patient is treated with LEAF-4L6715, a liposomal transcrocetin. The liposomal formulation allows for a gradual release of the free drug, thereby facilitating less frequent dosing.

Pharmacokinetic assessment will be carried out to identify an optimal dose and schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from the patient or patient's legal representative must be obtained prior to any procedures, as the likelihood of patients being able to provide consent is very limited
2. Patients must be ≥ 18 years old
3. Patient must have acute respiratory distress syndrome as defined, with a PaO2/FiO2 ratio of less than 200 mm Hg
4. Patient must be under artificial ventilation support (including patient under OptiflowTM Nasal High Flow device or an equivalent device)
5. Patient must have a life expectancy of at least 24 hours
6. Patients should have normal liver function as defined by ALT, AST and alkaline phosphate less than 3 ULN for the institution
7. Patient must have platelet count above >100,000 cells/mm3, hemoglobin > 8 g/dL and an absolute neutrophil count (ANC) of > 1000 cells/mm3
8. Patients requiring dialysis due to renal impairment in cohort 3

Exclusion Criteria:

1. Patient is enrolled in any other therapeutic clinical trial with the same endpoints. All observational studies or study with limited invasive methods (Pharmacokinetic studies, monitoring of virus charges studies, biological monitoring studies ….) are allowed
2. Patient is pregnant or breast-feeding
3. Patient has a known hypersensitivity to crocetins, LEAF-4L6715 or any of its excipients
4. Patients with hemoglobinopathy
5. Patients receiving extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
proportion of patients showing an increase of at least 25% of PaO2/FiO2 ratio | 24 hours

SECONDARY OUTCOMES:
proportion of patients with a PaO2/FiO2 ratio above 200 mm Hg | 24, 48 and 72 hours
all cause mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut de cancérologie Strasbourg Europe, Strasbourg

IPD SHARING:
Plan to Share IPD: No